CLINICAL TRIAL: NCT06693973
Title: An Early Clinical Study Evaluating the Safety and Efficacy of AcNK-Sup003 Cell Injection in the Treatment of Relapsed or Refractory B-cell Non-Hodgkin's Lymphoma
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: SupermAb (BeiJing) Biotech Co., Ltd (Unknown)
Responsible Party: Principal Investigator, MEI HENG, Wuhan Union Hospital, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Supermab01
Record Dates: First submitted 2024-11-13; First posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: B-cell Non-Hodgkin Lymphoma (B-NHL)
Keywords: CD19; CD20; NK cells
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- AcNK-Sup003 cell injection solution (Experimental): The AcNK technology has successfully achieved the direct, covalent, and directional conjugation of intact antibodies which includes the Fc domain to the surface of NK cells via a one-step enzymatic reaction. This novel approach yields a non-genetically modified NK cell that is conjugated with dual-targeting antibodies, referred to as AcNK. Specifically, AcNK-Sup003 cells are cryopreserved NK cells that have been conjugated with bispecific antibodies target both CD20 and CD19.
  Interventions: Drug: AcNK-Sup003 cell injection solution

INTERVENTIONS:
Drug: AcNK-Sup003 cell injection solution — The AcNK technology has successfully achieved the direct, covalent, and directional conjugation of intact antibodies which includes the Fc domain to the surface of NK cells via a one-step enzymatic reaction. This novel approach yields a non-genetically modified NK cell that is conjugated with dual-targeting antibodies, referred to as AcNK. Specifically, AcNK-Sup003 cells are cryopreserved NK cells that have been conjugated with bispecific antibodies target both CD20 and CD19.

SUMMARY:
The purpose of this study is to determine whether AcNK-Sup003 cell injection is safe and effective in the treatment of elapsed or refractory B-cell non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
The AcNK technology has successfully achieved the direct, covalent, and directional conjugation of intact antibodies which includes the Fc domain to the surface of NK cells via a one-step enzymatic reaction. This novel approach yields a non-genetically modified NK cell that is conjugated with dual-targeting antibodies, referred to as AcNK. Specifically, AcNK-Sup003 cells are cryopreserved NK cells that have been conjugated with bispecific antibodies target both CD20 and CD19. This clinical trial is an open-label, nonrandomized, investigator-initiated clinical trial to evaluate the safety, tolerability, pharmacokinetics, and efficacy of AcNK-Sup003 cell injection in patients with elapsed or refractory B-cell non-Hodgkin's lymphoma. The treatment cycle in this study is 28 days. A modified "3+3" design principle combined with accelerated titration is used, with three dose cohorts and one alternative dose cohort, each including 1 to 6 subjects (adjustments may be made based on the safety and efficacy results of enrolled subjects). The dose levels are: Dose Level 1: 3×10^8 AcNK-Sup003 cells, Dose Level 2: 1×10^9 AcNK-Sup003 cells, Dose Level 3: 3×10^9 AcNK-Sup003 cells, Dose Level 4 (alternative dose): 9×10^9 AcNK-Sup003 cells (with a flexibility range of ±20%). Treatments are administered up to three times from Day 0 to Day 14 of each cycle (recommended D0/D7/D14, the frequency of infusion per cycle may be adjusted by the investigator based on obtained PK data and the subject's actual situation).

ELIGIBILITY:
Inclusion Criteria:

1. Signed an informed consent form in writing and is able to comply with the visits and related procedures specified in the protocol.
2. Age ≥18 years old, with an expected survival of more than 3 months.
3. Confirmed by pathology to have CD20+ relapsed or refractory B-cell non-Hodgkin's lymphoma (according to the WHO 2016 lymphoma classification standards), including but not limited to diffuse large B-cell lymphoma, high-grade B-cell lymphoma, and grade 3b follicular lymphoma.
4. Relapsed or refractory disease, defined by one or more of the following:

   * Relapse, non-response, or progression after hematopoietic stem cell transplantation.
   * Disease stabilization but with a duration of ≤6 months after at least two cycles of second-line therapy (must have received CD20-targeted drugs [excluding CD20-negative tumors] and anthracycline drugs).
   * Disease progression or relapse after second-line therapy (must have received CD20-targeted drugs [excluding CD20-negative tumors] and anthracycline drugs).
5. ECOG performance status of 0-2.
6. Males with fertility potential and women of childbearing age must agree to use effective contraception from the time of signing the informed consent form until 6 months after the last administration of the study drug; women of childbearing age must have a negative pregnancy test at screening.
7. Lymphoma must have at least one measurable lesion according to the Lugano 2014 criteria, that is, lymph node lesions with a long diameter >15 mm or extranodal lesions with a long diameter >10 mm, and positive FDG-PET scan (5PS score of 4 or 5); lesions that have previously received radiotherapy are only considered measurable if there is clear evidence of radiographic disease progression after completion of radiotherapy.
8. Hematological parameters (within 7 days before testing without transfusion or hematopoietic growth factor treatment): Hemoglobin (Hb) ≥80 g/L, Absolute Neutrophil Count (ANC) ≥1×10^9/L, Platelet Count (PLT) ≥50×10^9/L.
9. Coagulation function: International Normalized Ratio (INR) ≤1.5×ULN, and Activated Partial Thromboplastin Time (APTT) ≤1.5×ULN (subjects on prophylactic anticoagulant therapy must have an INR between 2.0-3.0).
10. Hepatic, renal, and pulmonary function must meet the following requirements:

    1. Serum creatinine ≤1.5×ULN, or creatinine clearance ≥50 mL/min (estimated by the Cockcroft-Gault formula).
    2. Total bilirubin ≤1.5×ULN (≤3×ULN for subjects with liver lesions or Gilbert's syndrome).
    3. ALT and AST ≤3×ULN (≤5×ULN for subjects with liver lesions).
    4. Under indoor ventilation conditions and without oxygen supplementation, blood oxygen saturation is ≥92%.

Exclusion Criteria:

1. Primary central nervous system lymphoma, or active central nervous system involvement or symptoms of central involvement.
2. Accompanying active autoimmune diseases (e.g., systemic lupus erythematosus, rheumatoid arthritis, multiple sclerosis, Sjögren's syndrome, immune thrombocytopenia, etc.), uncontrolled multi-cavity effusions; presence of grade 2-4 acute graft-versus-host disease (GVHD) or moderate to severe chronic GVHD within 4 weeks before screening.
3. Severe cardiovascular and cerebrovascular history, including but not limited to:

   * Serious cardiac rhythm or conduction abnormalities, such as ventricular arrhythmias requiring clinical intervention, second- or third-degree atrioventricular block, etc.
   * Prolonged QT interval corrected by the Fridericia formula (QTcF), >450 ms for males; >470 ms for females.
   * Acute coronary syndrome, congestive heart failure, aortic dissection, stroke, or other grade 3 or higher cardiovascular and cerebrovascular events occurring within 6 months before screening.
   * Heart failure with a New York Heart Association (NYHA) functional classification of ≥II or left ventricular ejection fraction (LVEF) <50%.
   * Clinically uncontrollable hypertension, with systolic blood pressure still ≥160 mmHg and/or diastolic blood pressure ≥100 mmHg after standardized drug treatment.
4. Received autologous hematopoietic stem cell transplantation or other autologous cell therapy products within 3 months before lymphodepletion; received allogeneic hematopoietic stem cell transplantation or other allogeneic cell therapy products within 6 months before lymphodepletion; subjects who have undergone other organ transplants.
5. Received anti-tumor drug treatment or participated in other interventional clinical studies within 4 weeks before lymphodepletion or within 5 half-lives (whichever is shorter), including but not limited to chemotherapy drugs, small molecule targeted drugs, monoclonal antibodies, antibody-drug conjugates, etc.
6. Received live attenuated vaccine immunization or major surgery within 4 weeks before lymphodepletion, or subjects who require live attenuated vaccine immunization or major surgery during the study period.
7. Requires long-term (≥3 days) systemic corticosteroid treatment during the study period (dose ≥10 mg/day prednisone or equivalent corticosteroids), excluding inhaled or topical use; as determined by the investigator.
8. History of other malignant tumors (except for cervical carcinoma in situ, non-invasive basal cell or squamous cell skin cancer, or localized prostate cancer treated with radical therapy, and ductal carcinoma in situ after radical surgery) in the past or concurrently; suffering from severe diabetes or other severe underlying diseases.
9. Subjects with fungal, bacterial, viral, tuberculosis, or other infections requiring systemic anti-infective treatment within 14 days before lymphodepletion.
10. Positive for hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) with HBV DNA copies above the lower limit of detection; positive for hepatitis C virus (HCV) antibody with HCV RNA copies above the lower limit of detection; positive for human immunodeficiency virus (HIV) antibody; positive for syphilis spirochete antibody.
11. Has life-threatening hypersensitivity reactions or other intolerable conditions to the drugs used in the study, or severe allergic constitution.
12. Pregnant or breastfeeding women.
13. The investigator deems that the subject has other conditions that may affect compliance or is not suitable for participating in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2023-12-27 (Actual); Primary Completion 2026-01-13 (Estimated); Study Completion 2026-01-13 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicities (DLTs) | up to Day 28 post-infusion
serious adverse events (SAEs) | Through study completion, an average of 2 years
  The incidence, severity, and relationship to the study drug of all adverse events (AEs), including serious adverse events (SAEs). Adverse events would be assessed according to the Common Terminology Criteria for Adverse Events (CTCAE, Version 5.0)
Maximum tolerated dose | Through study completion, an average of 2 years

SECONDARY OUTCOMES:
Objective response rate (ORR) | up to 1 year after treatment of AcNK-Sup003
  Clinical efficacy would be evaluated according to 2014 Lugano criteria.
Duration of response (DOR) | Through study completion, an average of 2 years
  Clinical efficacy would be evaluated according to 2014 Lugano criteria.
Progression-free survival (PFS) | Through study completion, an average of 2 years
  PFS is defined as the interval between a subject's receipt of the first dose of AcNK-Sup003 cell infusion and the first assessment of disease progression or death.
Overall survival (OS) | Through study completion, an average of 2 years
  OS is defined as the interval between a subject's receipt of first AcNK-Sup003 cell infusion and death from any cause.
Cmax | up to Day 28 post-infusion
  Cmax is the peak expansion value of NK cells in peripheral blood.
Tmax | up to Day 28 post-infusion
  Tmax is the time to maximum concentration in peripheral blood.
AUC (0- day 28) | up to Day 28 post-infusion
  Area under the curve (0- day 28) refers to the area under curve of NK cell expansion between infusion and day 28 post infusion. They all reflect the pharmacokinetics.

OTHER OUTCOMES:
Changes in CD19 and/or CD20-positive B cells | Through study completion, an average of 2 years
Donor-specific HLA antibodies in the blood | Through study completion, an average of 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in cell therapy. Data or samples shared will be coded, with no PHI included. Approval of the request and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA).